CLINICAL TRIAL: NCT02272608
Title: Evaluation of Sleep Apnea Related Inflammation With CRP, ESR and Neutrophil toLymphocyte Ratio
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hakan Korkmaz, Assistant professor, Ordu University
Other Study IDs: Ordu University
Record Dates: First submitted 2014-10-12; First posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- control: patients WHO do not have sleep apnea
  Interventions: Other: Evaluation of Sleep Apnea Related Inflammation with CRP, ESR and Neutrophil toLymphocyte Ratio
- mild OSAS: mild apnea patients (AHI: 5-15)
  Interventions: Other: Evaluation of Sleep Apnea Related Inflammation with CRP, ESR and Neutrophil toLymphocyte Ratio
- moderate OSAS: moderate apnea patients (AHI: 16-30)
  Interventions: Other: Evaluation of Sleep Apnea Related Inflammation with CRP, ESR and Neutrophil toLymphocyte Ratio
- severe OSAS: severe OSAS patients (AHI: more than 30)
  Interventions: Other: Evaluation of Sleep Apnea Related Inflammation with CRP, ESR and Neutrophil toLymphocyte Ratio

INTERVENTIONS:
Other: Evaluation of Sleep Apnea Related Inflammation with CRP, ESR and Neutrophil toLymphocyte Ratio — CRP, ESR and Neutrophil toLymphocyte Ratio values of sleep apnea patients were evaluated with respect to apnea- hypopnea scores.

SUMMARY:
There is some evidence suggesting that OSA is associated with low level of systemic inflammation and oxidative stress. Low level systemic inflammation and subsequent vascular damage has been implicated as the underlying mechanism responsible for comorbidities. Detection of altered inflammatory markers in OSAS patients may predict the degree of nocturnal sleep disturbance and associated systemic inflammation and presence of comorbidities. Recently, novel inflammatory biomarkers, such as neutrophil to lymphocyte ratio (NLR) have been proposed as an indicator of systemic inflammation. To our knowledge, NLR has not been studied in OSAS. We conducted the present study to evaluate the association between OSAS and inflammatory markers CRP, ESR and NLR.

ELIGIBILITY:
Inclusion Criteria: Subjects who were referred for polysomnography (PSG) testing and performed the test were included Exclusion Criteria: Patients with malignancy, diabetes mellitus, dyslipidemia, cardiovascular disease or hypertension, chronic inflammatory processes, thyroid dysfunction, chronic hepatic disease, renal failure, any acute- subacute infectious disease within past 2 months, if data are incomplete such as blood sample testing results, if they were unable to perform complete PSG testing.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from sleep apnea and were referred to perform polysomnoraphy constituted the study groups. There were grouped into 4 according to apnea- hypopnea scores: control, mild apnea, moderate apnea and severe apnea.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of systemic inflammatory markers C-Reactive Protein, Erythrocyte Sedimentation Ratio and neutrophil to lymphocyte ratio in sleep apnea patients | After withdrawal of serum samples, patients were taken to sleep lab at the same day and polysomnography reports were evaluated 24 hours later